CLINICAL TRIAL: NCT01899417
Title: Analysis of Procedure-related Costs and Proposed Benefits of the ConforMIS iTotal® Cruciate Retaining Knee Replacement System Versus Standard Total Knee
Brief Title: Costs and Benefits of ConforMIS iTotal® Knee Replacement System Versus Standard Total Knee
Status: Completed | Type: Observational
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-001
Record Dates: First submitted 2013-07-09; First posted 2013-07-15 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis,Knee
Keywords: osteoarthritis; knee replacement; patient-specific; economics
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ConforMIS iTotal® Knee Replacement: knee joint replacement
  Interventions: Device: ConforMIS iTotal® Knee Replacement
- Standard Knee Replacements: knee joint replacement
  Interventions: Device: ConforMIS iTotal® Knee Replacement

INTERVENTIONS:
Device: ConforMIS iTotal® Knee Replacement — Patients that received a ConforMIS iTotal knee replacement versus other knee replacement devices.
  Other Names: Total knee replacement; arthoplasty; TKA; iTotal; Standard total knee device

SUMMARY:
The purpose of this study is to evaluate the costs and benefits of the ConforMIS iTotal® total knee replacement system versus standard total knee arthroplasty.

This study is designed to illustrate the difference in cost between standard total knee replacements and the ConforMIS iTotal at a single institution.

DETAILED DESCRIPTION:
STUDY DESIGN The study is a two-arm single-center, consecutively enrolled retrospective study. Patients enrolled will have previously received either an iTotal CR knee replacement or a standard total knee replacement. The study site will be located in the United States. A minimum of 100 with a maximum of 120 patients will be enrolled in each study arm for a maximum of 200 - 240 patients.

STUDY DURATION This study involves retrospective data collection of operative and peri-operative information to determine the cost impact of several surgical variables. The study will be complete when the retrospective data has been collected on up to 120 patients per arm.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received an iTotal or a standard total knee replacement
* Willingness to participate in the clinical study and to give informed consent, if necessary, as determined during IRB review
* >18 years of age

Exclusion Criteria:

* Participation in another clinical study that could confound results
* Patient is less than 3 months post-op

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a Total Knee Replacement performed by the Investigator and are at least 3 months post surgery.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Fixed and variable costs resulting from Total Knee Arthroplasty at 30 days post-op | 1 month
  Fixed and variable costs resulting from Total Knee Arthroplasty at 30 days post-op
Fixed and variable costs resulting from Total Knee Arthroplasty at 90 days post-op | 3 months
  Fixed and variable costs resulting from Total Knee Arthroplasty at 90 days post-op

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Martin, MD, Principal Investigator — JFK Medical Center
Locations (1):
- JFK Medical Center, Atlantis, Florida, United States

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Rougraff BT, Heck DA, Gibson AE. A comparison of tricompartmental and unicompartmental arthroplasty for the treatment of gonarthrosis. Clin Orthop Relat Res. 1991 Dec;(273):157-64. PMID 1959265
- [Background] Fitzpatrick C, FitzPatrick D, Lee J, Auger D. Statistical design of unicompartmental tibial implants and comparison with current devices. Knee. 2007 Mar;14(2):138-44. doi: 10.1016/j.knee.2006.11.005. Epub 2006 Dec 22. PMID 17188876
- [Background] Fitz W. Unicompartmental knee arthroplasty with use of novel patient-specific resurfacing implants and personalized jigs. J Bone Joint Surg Am. 2009 Feb;91 Suppl 1:69-76. doi: 10.2106/JBJS.H.01448. PMID 19182028
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035